CLINICAL TRIAL: NCT03194854
Title: Well-Being and Physical Activity Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Isaac Prilleltensky, Professor, School of Education and Human Development; Vice Provost, Office of Institutional Culture, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170541
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Health Promotion
Keywords: e-Health; self-efficacy theory; mixture modeling; mobile health; complier average causal effect estimation
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: The intervention group will be compared to a usual care (UC) control group on outcomes of self-efficacy, physical activity, and well-being. The intervention group will participate in online activities for 30 days while UC control group participants will be asked to conduct their lives as usual for the same 30 day period. Both groups will complete assessments during this time period. The UC group will be given access to the intervention for 30 days after all study participants have completed the three survey battery administrations.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants who have completed the full online T1 battery will be randomly assigned in real-time by the computer to either the intervention condition or the UC control condition. Randomization, group assignment, and assessments will be conducted solely by the computer program, so researchers will be blind to participant randomization, group assignment, and participant group identity during assessment times. With regard to group size and power, experience from our prior efficacy study of FFW indicates that for the current study, the computer program will use a 1:1 randomization algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fun For Wellness (FFW) (Experimental): Intervention participants will: 1) watch original videos with vignettes performed by professional actors; 2) read and/or watch mini-lectures that teach skills for behavior change; 3) engage in self-reflection exercises, 4) play original interactive games related to vignettes and mini-lectures; 5) interact with other FFW users via chat room functions and; 6) watch funny narrated video clips about well-being.
  Interventions: Behavioral: Fun For Wellness (FFW)
- Usual Care (UC) (No Intervention): The Usual Care (UC) group will conduct their lives as usual during the 30 day intervention period.

INTERVENTIONS:
Behavioral: Fun For Wellness (FFW) — FFW consists of videos, games, and content teaching 14 skills to support seven drivers of change that promote well-being in I COPPE domains. The drivers form the acronym BET I CAN, which stands for: Behaviors, Emotions, Thoughts, Interactions, Context, Awareness, and Next Steps. B teaches basics of habit formation, including antecedents, behaviors, and consequences and techniques like goal setting, behavior tracking and rewards. E teaches how to build positive emotions and cope with negative ones. T teaches lessons from cognitive behavioral therapy. I builds communication skills such as empathy, listening and assertiveness. C teaches how to create healthier environmental contexts. A aims to increase insight. N emphasizes the need to make plans and anticipate barriers.
  Arms: Fun For Wellness (FFW)

SUMMARY:
Fun For Wellness (FFW) is an online behavioral intervention designed to promote growth in well-being by providing capability-enhancing learning opportunities to participants. This study is a randomized controlled trial (RCT) designed to provide an initial evaluation of the effectiveness of FFW to increase well-being and physical activity in an obese adult population in the United States of America. The conceptual framework for the FFW intervention is guided by self-efficacy theory. The FFW intervention consists of participants engaging in BET I CAN challenges. BET I CAN is an acronym that stands for behaviors, emotions, thoughts, interactions, awareness, and next steps. The FFW intervention is conceptualized as exerting both a positive direct effect, and a positive indirect effect through self-efficacy (i.e., well-being self-efficacy), on well-being (i.e., subjective well-being and well-being actions).

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimates that 650 million adults are obese and that this number has tripled since 1975. To reduce adult obesity the WHO recommends that individuals limit energy intake from low quality food sources (e.g., highly processed foods high in fat), increase energy intake from high quality food sources (e.g., raw vegetables), and engage in regular physical activity (e.g., 150 minutes at moderate intensity per week). There is evidence, that well-designed cognitive-behavioral interventions can successfully promote physical activity in obese adults.

Insufficient physical activity in the general adult population is a global pandemic. At the individual-level, there is evidence that behavioral interventions designed to promote physical activity by focusing on personal psychological attributes (e.g., self-efficacy) can be effective. Delivering a physical activity intervention online has been shown to be an effective mode of delivery that also may allow for efficient scaling up of an intervention. Thus, a readily scalable online behavioral intervention that effectively promotes physical activity in obese adults may be useful in regard to responding to a global pandemic (i.e., physical inactivity) in an at-risk population (i.e., obese adults).

The conceptual framework for the Fun For Wellness intervention is based on self-efficacy theory. Over the past few decades, self-efficacy theory has been one of the most widely studied conceptual frameworks in sport and exercise psychology. FFW is an online behavioral intervention designed to promote growth in well-being by providing capability-enhancing learning opportunities to participants. For participants who comply with the intervention, some initial evidence has been provided for the efficacy of FFW to promote: well-being self-efficacy; interpersonal, community, psychological and economic subjective well-being; and, interpersonal and physical well-being actions.

A panel company will invite participants from their General Population member panel to go to the research webpage to be screened for the study. No more than six hundred obese adults (BMI ≥ 25.00 kg/m2) between 18 and 64 years old will be randomly assigned to the FFW or Usual Care (UC) group to achieve a 1:1 group (i.e. FFW:UC) assignment. Recruitment, eligibility verification and data collection will be conducted online. Data will be collected at baseline, 30 days and 60 days post-baseline. Instruments to measure demographic information, anthropometric characteristics, self-efficacy, physical activity, well-being, and health-related quality of life will be included in the battery. Data will be modeled under both an intent to treat approach and a complier average causal effect approach.

Primary outcomes are: well-being self-efficacy, subjective well-being and well-being actions.

Hypotheses for intervention compliers are:

1. The FFW intervention will exert a positive direct effect on well-being self-efficacy.
2. The FFW intervention will exert a positive direct effect on subjective well-being.
3. The FFW intervention will exert a positive direct effect on well-being actions.

Secondary outcomes are: well-being actions self-efficacy, physical activity self-efficacy, self-efficacy to regulate physical activity, and physical activity.

Hypotheses for intervention compliers are:

1. The FFW intervention will exert a positive direct effect on well-being actions self-efficacy.
2. The FFW intervention will exert a positive direct effect on physical activity self-efficacy.
3. The FFW intervention will exert a positive direct effect on self-efficacy to regulate physical activity.
4. The FFW intervention will exert a positive direct effect on physical activity.

Exploratory analyses will be conducted to examine possible relationships between the FFW intervention and health-related quality of life.

ELIGIBILITY:
There are seven eligibility criteria for participation in this study.

Inclusion Criteria:

* individual is at least 18 years old but not older than 64 years old
* individual has access to a technological device (e.g., computer) that can access the online intervention
* individual lives in the United States of America
* individual is not simultaneously enrolled in another program promoting either well-being or physical activity
* individual has a body mass index (BMI) ≥ 25.00 kg/m2

Exclusion Criteria:

* individual is less than 18 years old or older than 64 years old
* individual does not have access to a technological device (e.g., computer) that can access the online intervention
* individual does not live in the United States of America
* individual is simultaneously enrolled in another program promoting either well-being or physical activity
* individual has a body mass index (BMI) < 25.00

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2018-11-18 (Actual)

PRIMARY OUTCOMES:
Change in overall Well-Being Self-Efficacy (WBSE) Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on well-being self-efficacy.
Change in subjective well-being I COPPE Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on subjective well-being.
Change in I COPPE Actions Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on well-being actions

SECONDARY OUTCOMES:
Change in Well-Being Actions Self-Efficacy (WBASE) Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on well-being actions self-efficacy.
Change in Job-Related Physical Activity Self-Efficacy (J-R PASE) Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on job-related physical activity self-efficacy.
Change in Transportation-Related Physical Activity Self-Efficacy (T-R PASE) Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on transportation-related physical activity self-efficacy.
Change in Domestic-Related Physical Activity Self-Efficacy (D-R PASE) Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on domestic-related physical activity self-efficacy.
Change in Leisure-Related Physical Activity Self-Efficacy (L-R PASE) Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on leisure-related physical activity self-efficacy.
Change in Self-Efficacy to Regulate Physical Activity (SERPA) Scale scores between baseline and time 3. | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on self-efficacy to regulate physical activity.
Change in Long International Physical Activity Questionnaire (Long-IPAQ) scores between baseline and time 3 | baseline, 30 days, and 60 days
  The FFW intervention will exert a positive direct effect on physical activity.

OTHER OUTCOMES:
Relationships between FFW intervention and SF36v2 scores. | baseline, 30 days, and 60 days
  Exploratory analyses will be conducted to examine possible relationships between the FFW intervention and health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Prilleltensky, Ph.D., Principal Investigator — Professor, University of Miami, School of Education and Human Development; Vice Provost, Office of Institutional Culture; Nicholas D. Myers, Ph.D., Principal Investigator — Associate Professor, Michigan State University, Department of Kinesiology
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myers ND, Prilleltensky I, Lee S. Measuring stability and change in response patterns to a set of hierarchical scales in a randomized intervention study: an innovative application of latent transition analysis. J Behav Med. 2025 Aug 25. doi: 10.1007/s10865-025-00586-7. Online ahead of print. PMID 40853442
- [Derived] Myers ND, Brincks AM, Lee S. Direct and Indirect Causal Effects of an Individual Randomized Physical Activity-Promoting Intervention: A Substantive-Methodological Synergy. Meas Phys Educ Exerc Sci. 2025;29(1):24-42. doi: 10.1080/1091367x.2024.2392563. Epub 2024 Aug 19. PMID 40248477
- [Derived] Myers ND, Brincks AM, Lee S. Using Directed Acyclic Graphs (DAGs) to Determine if the Total Causal Effect of an Individual Randomized Physical Activity-Promoting Intervention is Identifiable. Meas Phys Educ Exerc Sci. 2024;28(3):267-282. doi: 10.1080/1091367x.2024.2318355. Epub 2024 Feb 19. PMID 39206182
- [Derived] Lee S, Myers ND, Bateman AG, Prilleltensky I, McMahon A, Brincks AM. Baseline self-efficacy predicts subsequent engagement behavior in an online physical activity intervention. Front Sports Act Living. 2024 Jul 3;6:1401206. doi: 10.3389/fspor.2024.1401206. eCollection 2024. PMID 39022641
- [Derived] Myers ND, Bateman AG, McMahon A, Prilleltensky I, Lee S, Prilleltensky O, Pfeiffer KA, Brincks AM. Measurement of Physical Activity Self-Efficacy in Adults With Obesity: A Latent Variable Approach to Explore Dimensionality, Temporal Invariance, and External Validity. J Sport Exerc Psychol. 2021 Nov 18;43(6):497-513. doi: 10.1123/jsep.2021-0040. PMID 34794118
- [Derived] Myers ND, Prilleltensky I, McMahon A, Brincks AM, Lee S, Prilleltensky O, Pfeiffer KA, Bateman AG. Mechanisms by Which the Fun for Wellness Intervention May Promote Subjective Well-Being in Adults with Obesity: a Reanalysis Using Baseline Target Moderation. Prev Sci. 2023 Feb;24(2):286-298. doi: 10.1007/s11121-021-01274-z. Epub 2021 Jun 25. PMID 34173135
- [Derived] Myers ND, McMahon A, Prilleltensky I, Lee S, Dietz S, Prilleltensky O, Pfeiffer KA, Bateman AG, Brincks AM. Effectiveness of the Fun for Wellness Web-Based Behavioral Intervention to Promote Physical Activity in Adults With Obesity (or Overweight): Randomized Controlled Trial. JMIR Form Res. 2020 Feb 21;4(2):e15919. doi: 10.2196/15919. PMID 32130110
- [Derived] Myers ND, Prilleltensky I, Lee S, Dietz S, Prilleltensky O, McMahon A, Pfeiffer KA, Ellithorpe ME, Brincks AM. Effectiveness of the fun for wellness online behavioral intervention to promote well-being and physical activity: protocol for a randomized controlled trial. BMC Public Health. 2019 Jun 13;19(1):737. doi: 10.1186/s12889-019-7089-2. PMID 31196052